CLINICAL TRIAL: NCT02618122
Title: A Multicenter, Prospective, oBservational Study to assEss the Clinical activitY and the Impact on symptOm Burden and patieNts' HRQoL of Treatment With trabecteDin in Advanced Soft Tissue Sarcomas in a Real World Setting in Greece. The 'beYOND-STS' Study
Brief Title: A Multicenter, Prospective, oBservational Study to assEss the Clinical activitY and Impact on symptOm Burden and patieNts' HRQoL of Treatment With trabecteDin in aSTS in a Real World Setting in Greece
Acronym: beYOND-STS
Status: Completed | Type: Observational
Sponsor: Genesis Pharma S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GEN-TRA-001
Record Dates: First submitted 2015-11-25; First posted 2015-12-01 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Advanced Soft Tissue Sarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This non-interventional study aims primarily at assessing the clinical effectiveness and the impact of the therapy on cancer-related symptoms and patients' HRQoL. In addition, it represents an attempt towards gaining experience on the routine use of trabectedin in daily clinical practice in a representative sample of Greek subjects with aSTS.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for inclusion in this study have to meet all of the following criteria:

* Adult outpatients (18 years and older) of either gender;
* Patients with a histologically confirmed diagnosis of advanced (locally advanced or metastatic) soft tissue sarcoma who have failed treatment with anthracyclines and ifosfamide or who are unsuited to receive these drugs;
* Patients for whom the decision to prescribe therapy with trabectedin (Yondelis®) according to the locally approved product's summary of product characteristics (SmPC) has already been taken prior to their enrolment in the study and is clearly separated from the physician's decision to include the patient in the current study;
* Patients must be able and willing to provide written informed consent and to comply with the requirements of this study protocol;
* Patients must have signed an informed consent document;
* Patients must be able to read, understand and complete the study specific questionnaires.

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from participation in this study:

* Patients who have received more than one cycle of trabectedin at the time of enrolment into the study;
* Patients that meet any of the contraindications to the administration of the study drug according to the approved SmPC;
* Patients who currently receive treatment with any investigational drug/device/intervention or have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) before the commencement of therapy with trabectedin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a histologically confirmed diagnosis of advanced (locally advanced or metastatic) soft tissue sarcoma who have failed treatment with anthracyclines and ifosfamide or who are unsuited to receive these drugs
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-08-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients that are alive and progression-free (as per the RECIST v1.1 criteria) 6 months after treatment commencement. | 6 months post-treatment onset
  The proportion of patients that are alive and progression-free (as per the RECIST v1.1 criteria) 6 months after treatment commencement

CONTACTS AND LOCATIONS:
Overall Officials: Kiki Karvounis, Study Director — GenesisPharma Medical Department
Locations (1):
- Thessaloniki, Thessaloniki, Greece